CLINICAL TRIAL: NCT01376076
Title: Evaluation of the Effects of Sequential Multiple-Dose Regimens of Cariprazine on Cardiac Repolarization in Patients With Schizophrenia
Brief Title: Effects of Cariprazine on Cardiac Repolarization in Patients With Schizophrenia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RGH-MD-02
Record Dates: First submitted 2011-06-16; First posted 2011-06-20 (Estimated); Last update posted 2012-02-08 (Estimated); Status verified 2012-02

CONDITIONS: Schizophrenia
Keywords: schizophrenia; QTc; cardiac repolarization
MeSH Terms: conditions — Schizophrenia | interventions — cariprazine; Risperidone; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Sequential, Multiple Dose, titration from 1.5mg to 18mg once daily dose of cariprazine
  Interventions: Drug: Cariprazine
- 2A (Placebo Comparator): Double blind placebo for Days 1-5, Moxifloxacin (400mg) on Day 6, Risperidone 4mg once daily Days 7-15, placebo Days 16-20, Risperidone Days 21-29, placebo Days 30-35
  Interventions: Drug: Risperidone/Moxifloxacin
- 2B (Placebo Comparator): Double blind placebo for Days 1-6, Risperidone 4mg once daily Days 7-15, placebo Days 16-20, Risperidone Days 21-29, placebo Days 30-34, Moxifloxacin (400mg) on Day 35
  Interventions: Drug: Risperidone/Moxifloxacin

INTERVENTIONS:
Drug: Cariprazine — Patients meeting all study eligibility criteria will be randomized to receive cariprazine (Group 1) 1.5 to 18 mg once daily, administered orally.
  Arms: 1
Drug: Risperidone/Moxifloxacin — Patients randomized to Group 2A will receive double blind placebo for Days 1-5, Moxifloxacin (400mg) on Day 6, Risperidone 4mg once daily Days 7-15, placebo Days 16-20, Risperidone Days 21-29, placebo Days 30-35.
  Arms: 2A
Drug: Risperidone/Moxifloxacin — Patients randomized to Group 2B will receive double blind placebo for Days 1-6, Risperidone 4mg once daily Days 7-15, placebo Days 16-20, Risperidone Days 21-29, placebo Days 30-34, Moxifloxacin (400mg) on Day 35.
  Arms: 2B

SUMMARY:
This study will evaluate the effects of sequential multiple dose regimens of cariprazine on cardiac repolarization in patients with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Men or women, age 18 to 50, inclusive
* Symptoms of schizophrenia or schizoaffective disorder first appearing a minimum of 1 year before screening
* Negative pregnancy test
* Normal physical examination results, vital signs, and clinical lab test results

Exclusion Criteria:

* Axis II disorder severe enough to interfere with the study
* Smoking more than 20 cigarettes a day
* History or presence of cardiovascular disorder
* Pregnant/breast-feeding and/or planning to become pregnant/breast-feed
* Imminent risk of injuring self or others or causing significant property damage

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 129 (Actual)
Dates: Start 2011-06; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Heart rate-corrected QT interval (QTc) | 35 days of double-blind treatment, up to 56 days total.
  The effects of a therapeutic dosage (9 mg/day) and a supratherapeutic dosage (18 mg/day) of cariprazine on cardiac repolarization as determined by heart-rate-corrected QT intervals will be assessed on Day 20 and Day 34, respectively. The assay sensitivity of moxifloxacin 400 mg/day will be assessed on Day 6 and Day 35.

CONTACTS AND LOCATIONS:
Overall Officials: Suneeta Ahuja, PhD, Study Director — Forest Laboratories
Locations (4):
- United States (4):
  - Forest Investigative Site 001, Glendale, California
  - Forest Investigative Site 004, Long Beach, California
  - Forest Investigative Site 002, Willingboro, New Jersey
  - Forest Investigative Site 003, Houston, Texas